CLINICAL TRIAL: NCT07070570
Title: HAKA: Routine Follow-up at 10 Years After Hip- or Knee Arthroplasty: Wasting Resources or Appropriate Healthcare?
Acronym: HAKA 10 years
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reinier Haga Orthopedisch Centrum (Other)
Collaborators: JointResearch (Other); Tergooi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OC-2024-011
Record Dates: First submitted 2025-07-14; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hip Arthroplasty, Total; Knee Arthroplasty, Total
Keywords: Routine follow-up; Check-up on demand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Follow-Up (RFU) (Other): Standard follow-up care with scheduled X-ray, clinical visit and questionnaires at 10 years after surgery
  Interventions: Other: Routine Follow-Up (RFU)
- Active Check-Up on Demand (ACOD) (Other): Follow-up care with X-ray, clinical visit and questionnaires at 10 years after surgery when requested by the patient or healthcare provider.
  Interventions: Other: Active Check-Up on Demand (ACOD)
- Passive Check-Up on Demand (PCOD) (Other): X-ray and clinical visit (without questionnaires) at 10 years after surgery when requested by the patient or healthcare provider.
  Interventions: Other: Passive Check-Up on Demand (PCOD)

INTERVENTIONS:
Other: Routine Follow-Up (RFU) — Standard follow-up care with scheduled X-ray, clinical visit and questionnaires at 10 years after surgery
  Arms: Routine Follow-Up (RFU)
Other: Active Check-Up on Demand (ACOD) — X-ray, clinical visit and questionnaires at 10 years after surgery when requested by the patient or healthcare provider.
  Arms: Active Check-Up on Demand (ACOD)
Other: Passive Check-Up on Demand (PCOD) — X-ray and clinical visit (without questionnaires) at 10 year when requested by the patient or healthcare provider.
  Arms: Passive Check-Up on Demand (PCOD)

SUMMARY:
After undergoing total hip or total knee arthroplasty, current guidelines recommend routine follow-up with an X-ray within 3 months and again at 1 year. Follow-up at 5 years (for hip arthroplasties) or every 5 years (for knee arthroplasties) is also considered worthwhile according to the guideline. However, these follow-up appointments require considerable time from patients, caregivers, and healthcare professionals, and it is unclear whether they are truly beneficial. It is possible that a single follow-up within 3 months is sufficient. This could potentially prevent over 100,000 unnecessary hospital visits per year, resulting in significant cost savings. If patients or healthcare providers have concerns, they can always request an additional follow-up.

The HAKA trial consists of three different work packages (WPs). This trial (WP2) investigates the 10-year follow-up, WP1 examines the 1-year follow-up, and WP3 is a qualitative study exploring the experiences and perceptions of patients and healthcare professionals. The aim of the HAKA trial is to safely reduce routine follow-up appointments after total hip or knee arthroplasty and to revise current clinical guidelines accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Underwent primary THA or TKA approximately 10 years ago
* Age 50 years or older at time of THA or TKA
* Capable and willing to complete questionnaires (when applicable)
* Understanding Dutch or English
* Willing to provide written informed consent in case the patient will complete questionnaires

Exclusion Criteria:

* Other indication for surgery than osteoarthritis
* Deceased
* Revision arthroplasty of hip or knee, except a conversion from unicompartmental knee arthroplasty to TKA or from hip hemiarthroplasty/resurfacing to THA
* Already participating in this study due to another hip or knee surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of complications | Assessed until 11 years after implantation
  The total number of post-operative complications per patient will be recorded.
Type of complications | Assessed until 11 years after implantation
  Complication types will be recorded and categorized (e.g., infection, periprosthetic fracture, loosening, malalignment, dislocation, prosthetic wear).
Healthcare consumption | Assessed at 10 years after implantation and then at 3 months, 6 months and 12 months.
  Healthcare consumption related to THA and TKA FU (number of X-rays and clinical visits)

SECONDARY OUTCOMES:
PROMIS Physical Function | Assessed at 10 and 11 years after implantation
  Patient-reported physical functioning will be assessed using the PROMIS® Physical Function Version 1.0, Short Form 10a. The short form consists of 10 items and is expressed by raw summed score ranging from 10 to 50, which can be converted to a T-score and SE. The T-score is a standardized score with a mean of 50 and a SD of 10. Higher T-scores indicate better physical functioning
Number of surgical interventions | Assessed until 11 years after implantation
  The total number of surgical re-interventions per patient related to the index procedure will be recorded.
Type of Surgical Interventions | Assessed until 11 years after implantation
  Types of surgical re-interventions will be recorded and categorized (e.g., DAIR, partial component exchange, full revision, irrigation and debridement without component retention).
Number of additional healthcare consumption | Assessed at 10 years after implantation and then at 3 months, 6 months and 12 months.
  Number of additional healthcare consumption related to THA or TKA FU (like clinical visit, telephone consultations, X-ray, CT scan, MRI scan, laboratory tests)
Type of additional healthcare consumption | Assessed at 10 years after implantation and then at 3 months, 6 months and 12 months.
  Type of additional healthcare consumption related to THA or TKA FU (like clinical visit, telephone consultations, X-ray, CT scan, MRI scan, laboratory tests)
Costs related to THA or TKA follow-up | Assessed at 10 years after implantation and then after at 3 months, 6 months and 12 months.
  Includes costs from electronic health records and additional patient questionnaires, covering hospital and non-hospital care.
Numeric Pain Rating Scale (NPRS) | Assessed at 10 and 11 years after implantation
  Patient-reported pain intensity, measured using a numeric scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores reflect more severe pain.
Numeric Satisfaction Rating Scale (NSRS) | Assessed at 10 and 11 years after implantation
  Numeric Rating Scale for satisfaction (NSRS) will be measured by a single question: "How satisfied are you with the results of the treatment?" The patient will answer this question with a NRS scale ranging from zero to ten. The higher the score, the better.
Health related quality of life (EQ-5D-5L) | Assessed at 10 years after implantation and then at 3 months, 6 months and 12 months
  Health-related quality of life is measured using the EQ-5D-5L questionnaire. The EQ-5D-5L index score ranges from -0.594 to 1.000, where 1.000 indicates full health, 0 represents death, and negative values represent health states worse than death. Higher scores indicate better health status

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier Haga Orthopedisch Centrum, Zoetermeer, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications (e.g., PROMs, healthcare consumption, complications) will be made available upon reasonable request. Metadata will be openly accessible with a persistent identifier.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available beginning 6 months after publication of the main results and will remain available for at least 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal and agree to a data use agreement will be granted access to de-identified IPD and selected supporting documents. Requests can be submitted to the corresponding author or data access contact. Access is conditional on approval by the study team.